CLINICAL TRIAL: NCT05101330
Title: Impact of Bilingual Prescription Medication Labels on Medication Adherence and Medication Management Self-Efficacy Among Elderly Singaporeans: A Pilot Study
Brief Title: Impact of Bilingual Prescription Medication Labels Among Elderly Singaporeans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was challenging, and no participants were recruited after 6 months despite minimizing these challenges. Therefore the study team has decided not to pursue this study any further.
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1
Record Dates: First submitted 2021-03-29; First posted 2021-11-01 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
Keywords: Medication adherence; Prescription Medication Labels; Bilingual prescription medication labels; Anti-diabetic drugs; Older adults; Medication management self-efficacy; Health literacy; Literacy; Anti-hypertensives; Glucose-lowering agent
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Medication Adherence; Literacy

STUDY DESIGN:
Intervention Model Description: We will recruit 40 patients who have just been given a new oral medication for a chronic disease. They will then be randomized (1:1) to either Pilot Trial A or Pilot Trial B.
  There will be 2 pilot versions of a 2-arm parallel-group RCT.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pilot Trial A, Usual Care arm (No Intervention): At recruitment, participants will be dispensed with new medication provided together with PMLs in English. After 2 weeks, data will be collected during a home visit and no changes will be made to the PMLs. After another 2 weeks, data will be collected and Rx Cap pill bottles will be retrieved.
- Pilot Trial A, Intervention arm (Experimental): At recruitment, participants will be dispensed new medication in Rx Cap pill bottles provided with PMLs in English. After 2 weeks, a home visit will be conducted, where the English PMLs will be switched out with bilingual PMLs. A final home visit will be done after another 2 weeks, and the labels will be switched back to the standard-issue PMLs issued by SGH, and the Rx Cap pill bottles will be retrieved.
  Interventions: Device: Bilingual prescription medication labels
- Pilot Trial B, Usual Care arm (No Intervention): At recruitment, participants will be dispensed new medication in Rx Cap pill bottles provided with PMLs in English. After 2 weeks, data will be collected and Rx Cap bottles will be retrieved.
- Pilot Trial B, Intervention arm (Experimental): At recruitment, participants will be dispensed new medication in Rx Cap pill bottles, provided with bilingual PMLs. After 2 weeks, data will be collected accordingly during the home visit and Rx Cap bottles will be retrieved. Bilingual labels will be removed and participants will resume usage of standard-issue SGH PMLs.
  Interventions: Device: Bilingual prescription medication labels

INTERVENTIONS:
Device: Bilingual prescription medication labels — The bilingual PML contains English and Chinese medication-related instructions for participants.
  Other Names: PMLs
  Arms: Pilot Trial A, Intervention arm; Pilot Trial B, Intervention arm

SUMMARY:
The proposed study aims to provide preliminary data that will enable the conduct of a larger Randomized Controlled Trial (RCT) on the impact of bilingual Prescription Medication Labels (PMLs) on 3 medication-related outcomes - medication adherence, medication management self-efficacy, and PML understanding.

DETAILED DESCRIPTION:
The investigators will randomize 40 patients to Pilot Trial A or Pilot Trial B. Those in Pilot Trial A will be further randomized to Bilingual PMLs (intervention arm) or English PMLs (usual care arm) at 2 weeks post-recruitment, after assessing baseline level of the 3 medication-related outcomes; trial outcomes: difference in change, from baseline to 2 weeks post-randomization, in the 3 medication-related outcomes between the 2 arms. Those in Pilot Trial B will be further randomized to Bilingual PMLs or English PMLs immediately post-recruitment; trial outcomes: difference, at 2 weeks post-randomization, in the 3 medication-related outcomes between the 2 arms. This formative study will (1) assess the feasibility of administering the intervention, (2) refine protocols for study participant recruitment, engagement and retention, and (3) gain experience with and refine measurement of the outcomes for evaluating the intervention. The conduct of 2 pilot trials will allow us to choose the optimal trial design and determine variability.

ELIGIBILITY:
Inclusion Criteria:

* Singapore citizen/permanent resident
* Aged 50 years and above
* Just received a new (i.e., not received before) oral medication for a chronic disease
* No moderate/severe cognitive impairment (5 or more correct responses on the Abbreviated Mental Test, AMT)
* Not deaf (self-reported)
* No binocular presenting near vision impairment (near visual acuity, with routinely used spectacles/lenses: at least 6/15 (0.40 logMAR) on the Landolt's C chart)
* Able to speak at least 1 of the 4 official languages;
* Unable to read in English but able to read another official language (as they will benefit the most from bilingual PMLs)
* Assessed as non-adherent

Exclusion Criteria:

- Patients who received, from the prescribing physician, a set of instructions for their new oral medication that does not match standard instructions (as the bilingual instructions for non-standard instructions would not be prepared for beforehand)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Estimated)

PRIMARY OUTCOMES:
Measuring change from Week 2 in Medication Adherence on the Adherence to Refills and Medications Scale (ARMS) at Week 4. (Pilot Trial A) | Week 2 and Week 4 of Pilot Trial A
  ARMS is a validated self-reported medication-adherence scale intended for patients with chronic diseases.
  Its 12 questions consist of 2 subscales - adherence to refilling prescriptions and adherence with taking medications. Each item is structured using the Likert scale, with the following response options and corresponding scores: "none" (score of 1), "some" (score of 2), "most" (score of 3 ), or "all of the time" (score of 4). The range of possible total scores is 12 to 48. Lower scores indicate better adherence.
Assessing Medication Adherence on the ARMS at Week 2. (Pilot Trial B) | Week 2 of Pilot Trial B
  ARMS is a validated self-reported medication-adherence scale intended for patients with chronic diseases.
  Its 12 questions consist of 2 subscales - adherence to refilling prescriptions and adherence with taking medications. Each item is structured using the Likert scale, with the following response options and corresponding scores: "none" (score of 1), "some" (score of 2), "most" (score of 3 ), or "all of the time" (score of 4). The range of possible total scores is 12 to 48. Lower scores indicate better adherence.
Measuring change from Week 2 in Medication Adherence using the MedTake Assessment at Week 4. (Pilot Trial A) | Week 2 and Week 4 of Pilot Trial A
  MedTake Assessment is a self-reported measure for pharmacy staff when providing pharmaceutical care services, assessing patient adherence and knowledge to dose, dosage, indication, food or water co-ingestion, and regimen. A composite score (0-100%); higher ~ better) summarizes patient's ability to take medicine safely.
Assessing Medication Adherence using the MedTake Assessment at Week 2 (Pilot Trial B) | Week 2 of Pilot Trial B
  MedTake Assessment is a self-reported measure for pharmacy staff when providing pharmaceutical care services, assessing patient adherence and knowledge to dose, dosage, indication, food or water co-ingestion, and regimen. A composite score (0-100%); higher ~ better) summarizes patient's ability to take medicine safely.
Measuring change from Week 2 in Medication Adherence via Pill Count at Week 4. (Pilot Trial A) | Week 2 and Week 4 of Pilot Trial A
  A pill count, in context of the new oral medication, will be done. % adherence = ((quantity dispensed)-(quantity remaining))/ ((prescribed number of pills per day) x (no. of days between dispensing date and interview))
Assessing Medication Adherence via Pill Count at Week 2. (Pilot Trial B) | Week 2 of Pilot Trial B
  A pill count, in context of the new oral medication, will be done. % adherence = ((quantity dispensed)-(quantity remaining))/ ((prescribed number of pills per day) x (no. of days between dispensing date and interview))
Measuring change from Week 2 in Medication Adherence based on Rx Cap openings at Week 4. (Pilot Trial A) | Week 2 and Week 4 of Pilot Trial A
  The Rx Cap Bluetooth smart cap automatically tracks medication usage every time it is opened. The data collected and stored within the Smart Cap will be imported at home visits with participants. Continuous (% adherence to prescribed regimen; 0-100%) and categorical variables (not at all; partially; fully) for medication adherence will be derived.
Assessing Medication Adherence based on Rx Cap openings at Week 2. (Pilot Trial B) | Week 2 of Pilot Trial B
  The Rx Cap Bluetooth smart cap automatically tracks medication usage every time it is opened. The data collected and stored within the Smart Cap will be imported at home visits with participants. Continuous (% adherence to prescribed regimen; 0-100%) and categorical variables (not at all; partially; fully) for medication adherence will be derived.
Measuring change from Week 2 in Medication management self-efficacy on the MUSE Scale at Week 4. (Pilot Trial A) | Week 2 and Week 4 of Pilot Trial A
  The 8-item Medication Understanding and Use Self-Efficacy Scale (MUSE), comprises of 2 subscales: (1) taking medication (4 items), and (2) learning about medication (4 items). Item scores (four-point Likert scale; strongly disagree (score 1), to, strongly agree (score=4)) will be summed for subscale (range: 4-16) and total scores (range: 8-32; higher score ~ greater level of medication management self-efficacy).
Measuring Medication management self-efficacy on the MUSE Scale at Week 2 (Pilot Trial B) | Week 2 of Pilot Trial B
  The 8-item Medication Understanding and Use Self-Efficacy Scale (MUSE), comprises of 2 subscales: (1) taking medication (4 items), and (2) learning about medication (4 items). Item scores (four-point Likert scale; strongly disagree (score 1), to, strongly agree (score=4)) will be summed for subscale (range: 4-16) and total scores (range: 8-32; higher score ~ greater level of medication management self-efficacy).
Measuring change from Week 2 in PML understanding at Week 4. (Pilot Trial A) | Week 2 and Week 4 of Pilot Trial A
  Respondents will be asked tailored questions (in their preferred language) specific to the instructions presented on their PML for the new oral medication.
Assessing PML understanding at Week 2. (Pilot Trial B) | Week 2 of Pilot Trial B
  Respondents will be asked tailored questions (in their preferred language) specific to the instructions presented on their PML for the new oral medication.

CONTACTS AND LOCATIONS:
Overall Officials: Giat Yeng Khee, PhD, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malhotra R, Bautista MAC, Muller AM, Aw S, Koh GCH, Theng YL, Hoskins SJ, Wong CH, Miao C, Lim WS, Malhotra C, Chan A. The Aging of a Young Nation: Population Aging in Singapore. Gerontologist. 2019 May 17;59(3):401-410. doi: 10.1093/geront/gny160. PMID 30517628
- [Background] Malhotra R, Bautista MAC, Tan NC, Tang WE, Tay S, Tan ASL, Pouliot A, Saffari SE, Chei CL, Vaillancourt R. Bilingual Text With or Without Pictograms Improves Elderly Singaporeans' Understanding of Prescription Medication Labels. Gerontologist. 2019 Mar 14;59(2):378-390. doi: 10.1093/geront/gnx169. PMID 29190378

DOCUMENTS (2):
  • Study Protocol (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT05101330/Prot_000.pdf
  • Informed Consent Form (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT05101330/ICF_001.pdf